CLINICAL TRIAL: NCT04956471
Title: Guideline - Based Nursing Plan for Dysphagia After Stroke: Current Status and Influencing Factors
Brief Title: Guideline - Based Nursing Plan for Dysphagia After Stroke
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019312
Record Dates: First submitted 2021-06-27; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospitalized patients with swallowing disorder after stroke,.
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — A sample method: convenience sampling, selecting A 3 armour hospital between September 2019 and January 2020 neurology hospital patients with swallowing disorder after stroke, about 15 cases.

SUMMARY:
Research purposes:1, investigate the nursing management is the head nurse for swallowing disorder after stroke care management status; Compared with the existing research, the difference between guidelines and evidence-based nursing plan and the analysis of the influencing factors.2, the investigation nursing personnel for swallowing disorder after stroke nursing implementation status; Compare the difference between its and department management requirements and to analyze its influencing factors.3 patients with swallowing disorder after stroke or their caregivers for swallowing disorder after stroke care needs of semi-structured interviews.

DETAILED DESCRIPTION:
Research purposes:1, investigate the nursing management is the head nurse for swallowing disorder after stroke care management status; Compared with the existing research, the difference between guidelines and evidence-based nursing plan and the analysis of the influencing factors.2, the investigation nursing personnel for swallowing disorder after stroke nursing implementation status; Compare the difference between its and department management requirements and to analyze its influencing factors.3 patients with swallowing disorder after stroke or their caregivers for swallowing disorder after stroke care needs of semi-structured interviews.Study design.This subject adopts the mixed methods research design, the three parts to complete. Research focuses on the 3 armour hospital for ten. The first part first USES the literature analysis method, systematic review of swallowing disorder after stroke related guidelines and research. According to the guidelines and involved in the study of swallowing disorder after stroke care issues related to design the head nurse questionnaire, then cross-sectional investigation understand swallowing disorder after stroke clinical nursing management present situation in our country. According to the regional distribution plans to choose 10 3 armour hospital survey, about 15 head nurse.The second part first USES the literature analysis method, systematic review of swallowing disorder after stroke related guidelines and research. According to the guidelines and involved in the study of brain 4 cross-sectional survey) 108%Understanding of the brain in our country。Hospital survey,About 250 nurses. The third part USES the qualitative research in the design of phenomenological research methods, through face-to-face semi-structured interviews, collect data, understand the needs of patients and their caregivers, guide the nursing measures of existing. Selection of founding of neurology ward patients as the research and interview object, about 20 cases need to sample.

ELIGIBILITY:
Inclusion criteria:

1. Cerebral apoplexy diagnosed by CT or MRI;
2. Drinking water from depression > grade 3;
3. Be clear and able to communicate;
4. Volunteer for the study.

Exclusion criteria:

1. If you have serious basic diseases such as cardiovascular and cerebrovascular diseases, you cannot cooperate with the examination.
2. The patient refused to accept the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 15 cases.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
1 swallowing disorder after stroke care management present situation investigation | One year after recruitment
  The first part of swallowing disorder after stroke care management present situation investigation; Investigation includes general information and management status. A data includes gender, age, working years, job position, cultural degree, whether to have participated in related training. Current conditions including room management specification, nurse training, swallowing dysfunction screening and evaluation management, nutrition, management of complications.

CONTACTS AND LOCATIONS:
Overall Officials: Baohua Li, Study Chair — Peking Yniversity Third Hospital Medical
Locations (1):
- Peking Yniversity Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No